CLINICAL TRIAL: NCT00238147
Title: Phase I Trial With Weekly Docetaxel, Capecitabine and Carboplatin as Induction Chemotherapy Followed by Concomitant Capecitabine and Radiotherapy in Patients With Locally Advanced Esophageal Cancer
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Patients Who Are Undergoing Surgery for Locally Advanced Esophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Masking: None | Purpose: Treatment
Other Study IDs: 6227; UWCC-UW-6227; AVENTIS-UW-03031; ROCHE-UW-03031; UW-03031; UWCC-04-2311-D-01; CDR0000445238 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Esophageal Cancer
Keywords: stage II esophageal cancer; stage III esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Capecitabine; Carboplatin; Docetaxel; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: capecitabine
Drug: carboplatin
Drug: docetaxel
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, carboplatin, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells. Capecitabine may also make tumor cells more sensitive to radiation therapy. Giving combination chemotherapy and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase I trial is studying the side effects and best dose of docetaxel when given together with carboplatin and capecitabine followed by chemoradiotherapy in treating patients who are undergoing surgery for locally advanced esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and dose-limiting toxicity of docetaxel when administered with carboplatin and capecitabine as neoadjuvant induction therapy in patients with locally advanced esophageal cancer.

Secondary

* Determine the qualitative and quantitative toxic effects of this regimen in these patients.
* Determine the clinical and pathological response in these patients treated with neoadjuvant induction therapy comprising docetaxel, carboplatin, and capecitabine followed by chemoradiotherapy with capecitabine.

OUTLINE: This is an open-label, dose-escalation study of docetaxel.

* Induction therapy: Patients receive docetaxel IV and carboplatin IV over 30-60 minutes on days 1, 8, and 15 and oral capecitabine twice daily on days 1-21. Treatment repeats every 28 days for 2 courses.

Cohorts of 3-6 patients receive escalating doses of docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Approximately 7 days after completion of induction therapy, patients proceed to chemoradiotherapy.

* Chemoradiotherapy: Patients receive oral capecitabine twice daily on days 1-42 and undergo radiotherapy once daily, 5 days a week, on days 1-40.
* Surgery: Approximately 4-8 weeks after completion of chemoradiotherapy, patients undergo surgery.

After completion of study treatment, patients are followed periodically for 5 years and then annually thereafter.

PROJECTED ACCRUAL: Approximately 18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed esophageal or gastroesophageal junction cancer

  * Locally advanced disease, meeting 1 of the following staging criteria:

    * T3, N0, M0 disease
    * Any T, N1, M0 disease
* Measurable or evaluable disease

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL

Hepatic

* Bilirubin normal
* Meets 1 of the following criteria:

  * Alkaline phosphatase (AP) normal AND AST/ALT ≤ 5 times upper limit of normal (ULN)
  * AP ≤ 2.5 times ULN AND AST/ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST/ALT normal

Renal

* Creatinine ≤ 2.0 mg/dL
* Creatinine clearance ≥ 80 mL/min

Cardiovascular

* No uncontrolled congestive heart failure
* No symptomatic coronary artery disease
* No uncontrolled arrhythmias
* No myocardial infarction within the past 12 months
* No other uncontrolled clinically significant cardiac disease

Gastrointestinal

* Able to swallow tablets
* Intact upper gastrointestinal tract
* No malabsorption syndrome

Immunologic

* No history of unanticipated severe reaction to fluoropyrimidine
* No known hypersensitivity to fluorouracil
* No severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No serious infection that requires continuous antibiotic therapy

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* No other prior or concurrent malignancy except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No history of seizures
* No history of serious psychiatric illness that would preclude study compliance or giving informed consent
* No peripheral neuropathy > grade 1

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy

Radiotherapy

* No prior radiotherapy

Other

* More than 28 days since prior investigational drugs
* No concurrent warfarin for active anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2004-09; Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sujata Rao, MD, Principal Investigator — Seattle Cancer Care Alliance
Locations (2):
- United States (2):
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington

REFERENCES:
- [Result] Rao S, Oelschlager BK, Koh WJ, et al.: Phase I trial with weekly docetaxel, capecitabine and carboplatin followed by concomitant capecitabine and radiotherapy in patients with locally advanced esophageal cancer. [Abstract] American Society of Clinical Oncology 2008 Gastrointestinal Cancers Symposium, 25-27 January 2008, Orlando, FL. A-123, 2008.